CLINICAL TRIAL: NCT04777448
Title: Optimised Management After Balloon Pulmonary Angioplasty in Patients With Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Optimized Management After Balloon Pulmonary Angioplasty in Chronic Thromboembolic Pulmonary Hypertension
Acronym: POpPART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EssaiClinique_POPPART
Record Dates: First submitted 2021-02-02; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic Thromboembolic Pulmonary Hypertension; Telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Simple physical activity advices will be given to the 27 patients of the control arm
- telerehabilitation (Experimental): Patients in the tele rehabilitation arm will perform 24 1h-telerehabilition sessions (dance, gym, cardio training, yoga, ...)
  Interventions: Procedure: telerehabilitation

INTERVENTIONS:
Procedure: telerehabilitation — 24 sessions (less Thant 1h hour each) of tele rehabilitation. Patients can choose among several activities (gym, dance, cardio training, ...)
  Arms: telerehabilitation

SUMMARY:
Balloon pulmonary angioplasty (BPA) is a new method of treatment for inoperable chronic thromboembolic pulmonary hypertension (CTEPH) or persistent CTEPH after surgery. BPA improves or even normalises hemodynamic parameters measured during a right heart catheterization. Nevertheless, the vast majority of patients retain dyspnea and impaired exercise capacity despite considerable hemodynamic improvements.

Pulmonary rehabilitation (RHB) can improve symptoms, quality of life and exercise capacity in patients with CTEPH. Unfortunately, access to RHB remains a concern in many countries. Tele-rehabilitation (tRHB) has been shown feasible and effective some cardiac or pulmonary diseases.

This randomized controlled study aims at comparing the effects of tRHB with the effects of simple advices regarding exercising in CTEPH patients with normalized or near-normalized pulmonary hemodynamics after BPA treatment.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a complication of pulmonary embolism leading to dyspnea, effort limitation and sometimes right heart failure and death. Balloon pulmonary angioplasty (BPA) is a new method of treatment for inoperable CTEPH or persistent CTEPH after surgery. BPA restores blood flow in the treated areas and improves or even normalises hemodynamic parameters measured during a right heart catheterization. Nevertheless, the vast majority of patients retain dyspnea and impaired exercise capacity after angioplasty procedures.

Exercise training has been demonstrated to alleviate exercise dyspnea and to improve exercise capacity in many chronic cardiopulmonary conditions. Pulmonary rehabilitation (RHB) can improve symptoms, quality of life and exercise capacity in patients with pulmonary vascular disease of different etiologies including CTEPH. Furthermore, RHB does not present any particular risk for CTEPH patients with normalized or near-normalized pulmonary hemodynamics. Unfortunately, access to RHB remains a concern in many countries. Tele-rehabilitation (tRHB) has been shown feasible and effective some cardiac or pulmonary diseases. Our hypothesis is that tRHB may also be effective in CTEPH patients with normalized or near-normalized pulmonary hemodynamics after BPA treatment.

This randomized controlled study aims at comparing the effects of tRHB with the effects of simple advices regarding exercising in CTEPH patients with normalized or near-normalized pulmonary hemodynamics after BPA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients who have undergone pulmonary angioplasty for CTEPH (group 4 of the international classification)
* Patients with a mean pulmonary artery pressure <= 30 mmHg and cardiac output > 2.5 L/min/m2 at the last angioplasty session
* Patients who had completed an incremental cardiopulmonary exercise test
* Patients affiliated to the French social security system
* Patients with signed informed consent

Exclusion Criteria:

* Patients unable to complete an incremental cardiopulmonary exercise test
* Patients unable to complete a 6-minutes walking test, 3-minutes chair raising test and a rehabilitation
* Patient unable, for technical or any other reason, to connect via the Internet for remote monitoring and/or telerehabilitation
* Patient for whom a refusal to participate in a rehabilitation programme is anticipated
* Patient who has participated in a rehabilitation programme in the 6 months prior to the date of inclusion
* Patients referred to in Articles L1121-5 to L1121-8 of the CSP (pregnant women, parturients, nursing mothers, persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care and adults subject to a legal protection measure or unable to express their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Difference of endurance time on cycloergometer | At inclusion and after 3 months
  Expressed in seconds and calculated as follow: endurance time after 3 months - endurance time at inclusion The two tests are performed at 80% of the maximum power reached during a maximum incremental effort test (performed before inclusion)

SECONDARY OUTCOMES:
6-minutes walking test (6MWT) | At inclusion and at Month 3
  Distance walked in 6-min (in meters)
3-minutes chair rise test (3-CRT) | At inclusion and at Month 3
  Number of rises during 3-CRT (n)
SF-36 | At inclusion and at Month 3
  Physical dimensions of the SF-36 questionnaire
Dyspnea (NYHA scale) | At inclusion, at Month 1, Month 2 and Month 3
  Either I, II, III or IV
Telerehabilitation | Through study completion, an average of 3 months
  Total number of sessions achieved
St George Respiratory Questionnaire (SGRQ) | At inclusion and at Month 3
  Total SGRQ score
Dyspnea (mMRC score) | At inclusion, at Month 1, Month 2 and Month 3
  Either 0, 1, 2, 3 or 4

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Degano, MD, PhD, Principal Investigator — CHU Grenoble Alpes

IPD SHARING:
Plan to Share IPD: No